CLINICAL TRIAL: NCT02593591
Title: Clinical Sequencing Project for Metastatic Cancer Patients for Personalized Cancer Clinic.
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung tae Kim, MD,PhD,Division of hematology-oncology,Department of medicine, Samsung Medical Center
Other Study IDs: 2015-10-063
Record Dates: First submitted 2015-10-26; First posted 2015-11-02 (Estimated); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomarker group: Advanced cancer undergoing genomic profiling

SUMMARY:
The next generation of personalized medical treatment according to the type of personal genetic information are evolving rapidly. The genome analysis needs systematic infra and database based on personal genetic information. Therefore, a big data of genome-clinical information is important.

To determine the feasibility of the use of tumor's molecular profiling and targeted therapies in the treatment of advanced cancer and to determine the clinical outcome(Response rate,PFS, duration of response and overall survival )of patients with advanced cancer, the investigators are going to take a tumor tissue of patients and process molecular profiling and receive molecular profile directed treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 19 years of age.
2. Subject has a histologically or cytologically confirmed diagnosis of Colorectal cancer.
3. Prior treatment with anti-PDL1 antibody or immune check point inhibitor or ramucirumab therapy in the First-line or maintenance setting is allowed
4. They must have refractory or progressive disease for which there is no further curative therapy available.
5. Be willing to provide fresh tissue for biomarker analysis, and, based on the adequacy of the tissue sample quality for assessment of biomarker status.
6. Must have a life expectancy of 3 months or more
7. Written and voluntary informed consent understood, signed and dated.

Exclusion Criteria:

1. Patients who do not have enough tissue for acquisition

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with treatment-refractory malignancy
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Response rate | 1 year

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
Duration of response | 1 year
overall survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, Korea, Republic of, South Korea